CLINICAL TRIAL: NCT06521554
Title: A Phase 1a/1b Study of the Selective Tyrosine Kinase Inhibitor NVL-330 in Patients With Advanced or Metastatic HER2-altered NSCLC (HEROEX-1)
Brief Title: A Study of NVL-330 in Patients With Advanced or Metastatic HER2-altered NSCLC (HEROEX-1)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvalent Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NVL-330-01
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a dose escalation (Experimental): NVL-330 oral daily dosing
  Interventions: Drug: NVL-330
- Phase 1b dose expansion (Experimental): NVL-330 oral daily dosing
  Interventions: Drug: NVL-330

INTERVENTIONS:
Drug: NVL-330 — Oral Tablet of NVL-330

SUMMARY:
Phase 1a/1b dose escalation and expansion study designed to evaluate the safety and tolerability of NVL-330, determine the recommended Phase 2 dose (RP2D), and evaluate the antitumor activity in patients with advanced or metastatic HER2-altered NSCLC.

Phase 1a dose escalation is designed to assess the safety and tolerability of NVL-330 and to select the candidate RP2D(s) and, if applicable, the MTD.

Phase 1b expansion is designed to further evaluate the overall safety and tolerability of the candidate RP2D(s) of NVL-330 and to determine the RP2D of NVL-330 in patients with advanced or metastatic HER2 mutant NSCLC.

DETAILED DESCRIPTION:
The planned Phase 1a/1b first-in-human study is designed as a two-part clinical trial to investigate NVL-330 in pre-treated patients with advanced or metastatic HER2-altered NSCLC. The dose escalation phase of the trial is designed to enroll a set number of patients per cohort at protocol defined dose levels.

After the initial patients are treated at a given dose level and monitored for at least 28 days, available data will be reviewed, and initiation of the next dosing group will proceed with consideration given to the overall safety profile.

The expansion phase of the trial is designed to further evaluate safety and activity and to confirm the RP2D(s).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically confirmed locally advanced or metastatic NSCLC
3. Documented HER2 status as follows:

   1. Phase 1a: Documented oncogenic HER2 mutation such as HER2 exon20 insertion mutations or single nucleotide variants or HER2 amplification.
   2. Phase 1b: Documented oncogenic HER2 mutation.
4. Identification of lesions as follows:

   1. Phase 1a: Must have evaluable disease (target or nontarget) according to RECIST 1.1.
   2. Phase 1b: Must have measurable disease, defined as ≥ 1 radiologically measurable target lesion according to RECIST 1.1.
5. Adequate organ function and bone marrow reserve

Exclusion Criteria:

1. Patient's cancer has known oncogenic driver alteration other than HER2
2. Known allergy/hypersensitivity to excipients of NVL-330
3. Major surgery within 4 weeks of the first dose of study drug
4. Ongoing or recent anticancer therapy
5. Actively receiving systemic treatment or direct medical intervention on another therapeutic clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | As determined by incidence of DLTs during the first 28 days of treatment (ie, Cycle 1)
  To determine up to 2 RP2D Candidates
Maximum Tolerated Dose (MTD) | As determined by incidence of DLTs during the first 28 days of treatment (ie, Cycle 1)
  If applicable, to determine the MTD
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) | First dose of study drug through 30 days after the last dose of study drug
  Number of participants with TEAEs as assessed by CTCAE, v5.0

SECONDARY OUTCOMES:
Effect of Food on Maximum Plasma Concentration (Cmax) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the effect of food on maximum plasma concentration (Cmax) of NVL-330
Effect of Food on Area Under the Curve from Time 0 to 24 (AUC0-24) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the effect of food on area under the curve from time 0 to 24 of NVL-330
Effect of Food on Area Under the Curve from Time 0 to Infinity (AUCinf) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the effect of food on area under the curve from time 0 to infinity of NVL-330
Effect of Food on Time of Maximum Concentration (Tmax) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the effect of food on time of maximum concentration of NVL-330
Maximum plasma concentration (Cmax) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the maximum plasma concentration (Cmax) of NVL-330
Maximum plasma concentration (Cmax- dose normalized) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the maximum plasma concentration (Cmax-dose normalized) of NVL-330
Plasma concentration at the end of the dosing interval (Ctau) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the plasma concentration at the end of the dosing interval (Ctau) of NVL-330
Plasma concentration 24 hours post-dose (C24) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the plasma concentration 24 hours post-dose (C24) of NVL-330
Average plasma concentration (Cavg) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the average plasma concentration (Cavg) of NVL-330
Time of maximum concentration (Tmax) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the time of maximum concentration (Tmax) of NVL-330
Area Under the Curve at the End of the Dosing Interval (AUCtau) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve at the end of the dosing interval (AUCtau) of NVL-330
Area Under the Curve at the End of the Dosing Interval (AUCtau - dose normalized) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve at the end of the dosing interval (AUCtau - dose normalized) of NVL-330
Area Under the Curve From Time 0 to 24 (AUC0-24) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to 24 (AUC0-24) of NVL-330
Area Under the Curve From Time 0 to 24 (AUC0-24 - dose normalized) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to 24 (AUC0-24 - dose normalized) of NVL-330
Area Under the Curve From Time 0 to Infinity (AUCinf) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to infinity (AUCinf) of NVL-330
Area Under the Curve From Time 0 to Infinity (AUCinf - dose normalized) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to infinity (AUCinf - dose normalized) of NVL-330
Oral clearance (CL/F) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the oral clearance (CL/F) of NVL-330
Volume of Distribution (Vz/F) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the volume of distribution (Vz/F) of NVL-330
Accumulation Ratio of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the ratio of accumulation of NVL-330
Half-life (t1/2) of NVL-330 | Pre-dose and up to 24 hours post-dose
  To determine the half-life (t1/2) of NVL-330
Objective Response Rate (ORR) | 2 -3 years after first patient dosed
  Objective Response Rate (ORR) as determined by RECIST 1.1 criteria
Duration of Response (DOR) | 2 to 3 years after first patient dosed
  Time from first investigator-assessed response to radiographic disease progression or death
Intracranial Objective Response Rate (IC-ORR) | 2 to 3 years after first patient dosed
  The proportion of patients with a confirmed intracranial response (IC-CR or IC-PR)
Intracranial Duration of Response (IC-DOR) | 2 to 3 years after first patient dosed
  The time from first investigator-assessed intracranial response to radiographic intracranial disease progression or death
Time to Response (TTR) | Approximately 3 years
  The time from first dose to first confirmed radiographic response

CONTACTS AND LOCATIONS:
Overall Officials: Steve Margossian, MD PhD, Study Director — Nuvalent Inc.
Locations (21):
- United States (17):
  - City of Hope - Lennar, Irvine, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Institute, Stanford, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OSU Brain and Spine Hospital, Columbus, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - North Shore Health Hub, Saint Leonards, New South Wales
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Center - University Health Network, Toronto, Ontario